CLINICAL TRIAL: NCT01022853
Title: An Open Label Phase I Dose Escalation Trial of Intravenous BI 6727 in Combination With Oral BIBF 1120 in Patients With Advanced Solid Tumours With Repeated Administration in Patients With Clinical Benefit
Brief Title: Combination of BI6727 (Volasertib) and BIBF1120 in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1230.7; 2008-008304-41 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2017-10

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — BI 6727; nintedanib

ARMS (1):
- BIBF 1120 and BI 6727 (Experimental): Finding Maximum Tolerated Dose of BI 6727 in combination with BIBF 1120
  Interventions: Drug: BI 6727; Drug: BIBF 1120

INTERVENTIONS:
Drug: BI 6727 — intravenous each 21 days
Drug: BIBF 1120 — oral continuously

SUMMARY:
The primary objective of the current study is to investigate the Maximum Tolerated Dose (MTD) in terms of safety and tolerability of BI 6727 in combination with fixed dose BIBF 1120, in patients with advanced or metastatic solid tumours.

ELIGIBILITY:
Inclusion criteria:

1. Patients with confirmed diagnosis of advanced, non resectable and/or metastatic solid tumours, who have failed conventional treatment, and for whom no therapy of proven efficacy exists, or who are not amenable to established forms of treatment
2. Age > or = 18 years
3. European Cooperative Oncology Group performance status < or = 2
4. Written informed consent in accordance with International Conference on Harmonization -Good Clinical Practice (ICH-GCP) and local legislation
5. Recovery from Common Terminology Criteria for Adverse Events grade 2-4 therapy-related toxicities from previous systemic anti-cancer therapies or radiotherapy (except alopecia)

Exclusion criteria:

1. Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the trial
2. Known hypersensitivity to the trial drugs or their excipients
3. Treatment with any other investigational drug or participation in any other interventional trial within 28 days before first administration of trial drug (BIBF 1120) or concomitantly with this trial
4. Systemic anti-cancer therapy or radiotherapy within 28 days before start of therapy or concomitantly with this trial. The restriction does not apply to steroids and bisphosphonates
5. Active infectious disease infection or HIV I/II
6. Other malignancy currently requiring another anti-cancer therapy
7. Clinical evidence of symptomatic progressive brain or leptomeningeal disease during the past 6 months
8. Known inherited predisposition to bleeding or thrombosis
9. Radiographic evidence of cavitary or necrotic tumours
10. History of clinically significant haemoptysis within the past 3 months
11. Centrally located tumours with radiographic evidence (Computed Tomography or Magnetic Resonance Imaging) of local invasion of major blood vessels
12. Absolute Neutrophil Count (ANC) less than 1.5 x 1000000000/L
13. Platelets Count (PLT) less than 100 x 1000000000/L
14. Total bilirubin > upper limit of normal (ULN)
15. Alaninaminotransferase (ALT) and/or Aspartateaminotransferase (AST) >= 1.5 x ULN (in case of liver metastases: ALT and AST >= 2.5 x ULN)
16. Serum creatinine > 1.5 mg/dl
17. Major injuries and/or surgery or bone fracture within 28 days before first administration of trial drug (BIBF 1120), or planned surgical procedures during the trial period
18. Known history of clinically relevant QT prolongation (e.g. long QT syndrome)
19. History of severe haemorrhagic or thromboembolic event in the past 6 months (excluding central venous catheter thrombosis and peripheral deep vein thrombosis)
20. Therapeutic anticoagulation (except low dose heparin and/or heparin flush as needed for maintenance of an indwelling intravenous device) or antiplatelet therapy (except for chronic low-dose therapy with acetylsalicylic acid < or = 325mg per day)
21. Active alcohol or drug abuse
22. Women and men who are sexually active and unwilling to use a medically acceptable method of contraception during the trial
23. Pregnancy or breast-feeding
24. Patients unable to comply with the protocol
25. Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Italy (2):
  - 1230.7.39002 Boehringer Ingelheim Investigational Site, Ancona
  - 1230.7.39001 Boehringer Ingelheim Investigational Site, Milan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An uncontrolled, open-label, dose escalation study in cohorts of patients following the '3+3 design with de-escalation'. After entering the study, cohorts of patients were sequentially allocated to the dose levels.
Pre-assignment Details: Beginning after the first cycle of treatment, intra-patient dose escalations were allowed and could be repeated after every cycle. Intra-patient dose escalation was not allowed after the maximum tolerated dose (MTD) was determined.
Groups:
- 100 mg Volasertib + 200 mg Nintedanib: Course 1 comprised of 28 days because of a 7-day run-in period for nintedanib (200 mg twice daily). The treatment with nintedanib started on Day 1 of Course 1 and continued until the end of the course. 100 mg volasertib was infused on Day 8 of Course 1; no nintedanib was to be taken on that day.
  Course 2 and subsequent courses comprised 21 days. Volasertib was infused on Day 1 and continuous nintedanib administration re-started on Day 2.
- 200 mg Volasertib + 200 mg Nintedanib: Course 1 comprised of 28 days because of a 7-day run-in period for nintedanib (200 mg twice daily). The treatment with nintedanib started on Day 1 of Course 1 and continued until the end of the course. 200 mg volasertib was infused on Day 8 of Course 1; no nintedanib was to be taken on that day.
  Course 2 and subsequent courses comprised 21 days. Volasertib was infused on Day 1 and continuous nintedanib administration re-started on Day 2.
- 300 mg Volasertib + 200 mg Nintedanib: Course 1 comprised of 28 days because of a 7-day run-in period for nintedanib (200 mg twice daily). The treatment with nintedanib started on Day 1 of Course 1 and continued until the end of the course. 300 mg volasertib was infused on Day 8 of Course 1; no nintedanib was to be taken on that day.
  Course 2 and subsequent courses comprised 21 days. Volasertib was infused on Day 1 and continuous nintedanib administration re-started on Day 2.
- 350 mg Volasertib + 200 mg Nintedanib: Course 1 comprised of 28 days because of a 7-day run-in period for nintedanib (200 mg twice daily). The treatment with nintedanib started on Day 1 of Course 1 and continued until the end of the course. 350 mg volasertib was infused on Day 8 of Course 1; no nintedanib was to be taken on that day.
  Course 2 and subsequent courses comprised 21 days. Volasertib was infused on Day 1 and continuous nintedanib administration re-started on Day 2.
- 400 mg Volasertib + 200 mg Nintedanib: Course 1 comprised of 28 days because of a 7-day run-in period for nintedanib (200 mg twice daily). The treatment with nintedanib started on Day 1 of Course 1 and continued until the end of the course. 400 mg volasertib was infused on Day 8 of Course 1; no nintedanib was to be taken on that day.
Period: Overall Study
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib | 400 mg Volasertib + 200 mg Nintedanib
Started | 3 (entered and treated) | 4 (entered and treated) | 13 (entered and treated) | 8 (entered and treated) | 2 (entered and treated)
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 4 | 13 | 8 | 2
Not completed — Progressive disease | 2 | 3 | 11 | 7 | 1
Not completed — Dose-limiting toxicity | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 0
Not completed — Other not stated above | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set - All patients who received ≥1 dose of study medication were included in the treated set.
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib | 400 mg Volasertib + 200 mg Nintedanib | Total
Number analyzed (Participants) | 3 | 4 | 13 | 8 | 2 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (9.2) | 60.0 (7.1) | 57.5 (8.8) | 53.1 (12.9) | 59.0 (5.7) | 56.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 7 | 2 | 1 | 12
  Male | 2 | 3 | 6 | 6 | 1 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in the First Cycle for the Determination of the Maximum Tolerated Dose (MTD).
Description: DLT was defined as:
  1. Drug-related CTCAE (Common Terminology Criteria for Adverse Events) grade 3 or 4 non-haematological toxicity (except untreated vomiting, untreated nausea, or untreated diarrhoea) or
  2. Drug-related CTCAE grade 4 neutropenia for 7 or more days and/or complicated by infection or
  3. CTCAE grade 4 thrombocytopenia
Time Frame: 28 days
Population: Treated set. All patients who received ≥1 dose of study medication were included in the treated set.
Measure: Number; unit: participants
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib | 400 mg Volasertib + 200 mg Nintedanib
Number analyzed (Participants) | 3 | 4 | 13 | 8 | 2
participants | 0 | 0 | 3 | 2 | 2

2. Secondary Outcome: Number of Participants With Drug Related Adverse Events
Description: Number of participants with investigator-defined drug related adverse events.
Time Frame: From first study drug administration until 28 days after the last administration of any study medication, up to 485 days
Population: Treated Set.
Measure: Number; unit: participants
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib | 400 mg Volasertib + 200 mg Nintedanib
Number analyzed (Participants) | 3 | 4 | 13 | 8 | 2
participants | 3 | 3 | 12 | 7 | 2

3. Secondary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Number of participants with dose limiting toxicities (DLTs).
  DLT was defined as:
  1. Drug-related CTCAE grade 3 or 4 non-haematological toxicity (except untreated vomiting, untreated nausea, or untreated diarrhoea) or
  2. Drug-related CTCAE grade 4 neutropenia for 7 or more days and/or complicated by infection or
  3. CTCAE grade 4 thrombocytopenia
Time Frame: as for outcome 2
Population: Treated Set.
Measure: Number; unit: participants
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib | 400 mg Volasertib + 200 mg Nintedanib
Number analyzed (Participants) | 3 | 4 | 13 | 8 | 2
participants | 0 | 1 | 6 | 2 | 2

4. Secondary Outcome: Cmax of Volasertib
Description: Maximum measured concentration (Cmax) in plasma of Volasertib in Cycle 1.
Time Frame: 0:05 h before start of Volasertib infusion and 1:00, 2:00, 3:00, 4:00, 8:00 and 24 h after start of Volasertib infusion
Population: Pharmacokinetic (PK) analysis set. The PK analysis set included all patients who took at least 1 dose of study medication and provided at least 1 blood sample following drug administration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib | 400 mg Volasertib + 200 mg Nintedanib
Number analyzed (Participants) | 3 | 4 | 12 | 6 | 2
ng/mL | 164 (77.6) | 409 (23.3) | 532 (33.3) | 534 (25.5) | 1210 (54.1)

5. Secondary Outcome: CL of Volasertib
Description: Total plasma Clearance (CL) of Volasertib in Cycle 1.
Time Frame: 0:05 h before start of Volasertib infusion and 1:00, 2:00, 3:00, 4:00, 8:00 and 24 h after start of Volasertib infusion
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib | 400 mg Volasertib + 200 mg Nintedanib
Number analyzed (Participants) | 3 | 4 | 10 | 5 | 2
mL/min | 720 (19.30) | 685 (4.22) | 792 (34.2) | 849 (29.3) | 589 (18.3)

6. Secondary Outcome: Vss of Volasertib
Description: Volume of distribution at steady state (Vss) of Volasertib in Cycle 1.
Time Frame: 0:05 h before start of Volasertib infusion and 1:00, 2:00, 3:00, 4:00, 8:00 and 24 h after start of Volasertib infusion
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib | 400 mg Volasertib + 200 mg Nintedanib
Number analyzed (Participants) | 3 | 4 | 10 | 5 | 2
L | 5710 (39.9) | 5590 (6.53) | 5010 (34.7) | 6080 (21.2) | 2710 (87.3)

7. Secondary Outcome: Cmax of Nintedanib
Description: Maximum measured concentration (Cmax) of Nintedanib in Cycle 1.
  400 mg Volasertib + 200 mg Nintedanib group is not displayed due to data only being available for one patient.
Time Frame: 5 min before Nintedanib administration in the morning and 1:00, 2:00, 3:00, 4:00, 6:00 h after administration on Day 9
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib
Number analyzed (Participants) | 3 | 4 | 6 | 4
ng/mL | 22.5 (58.0) | 30.2 (66.2) | 36.7 (53.3) | 34.2 (53.8)

8. Secondary Outcome: AUC(0-6h) of Nintedanib
Description: Area under the concentration-time curve (AUC) of Nintedanib over the time interval 0 to 6 hours in Cycle 1.
  400 mg Volasertib + 200 mg Nintedanib group is not displayed due to data only being available for one patient.
Time Frame: 5 min before Nintedanib administration in the morning and 1:00, 2:00, 3:00, 4:00, 6:00 h after administration on Day 9
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib
Number analyzed (Participants) | 3 | 4 | 6 | 4
ng*h/mL | 69.5 (29.9) | 104.0 (59.4) | 135.0 (48.8) | 121.0 (51.0)

9. Secondary Outcome: Tmax of Nintedanib
Description: Time from dosing to the maximum measured concentration, Cmax, of Nintedanib (tmax) in Cycle 1.
  400 mg Volasertib + 200 mg Nintedanib group is not displayed due to data only being available for one patient.
Time Frame: 5 min before Nintedanib administration in the morning and 1:00, 2:00, 3:00, 4:00, 6:00 h after administration on Day 9
Population: PK analysis set.
Measure: Median (Full Range); unit: h
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib
Number analyzed (Participants) | 3 | 4 | 6 | 4
h | 3.00 [3.00 to 3.00] | 1.88 [1.00 to 2.75] | 2.42 [1.00 to 3.00] | 2.00 [1.00 to 6.00]

10. Secondary Outcome: Number of Patients With Best Overall Response
Description: Best overall response based on response evaluation criteria in solid tumors (RECIST) version 1.1. Best overall response is defined as the best overall response (complete response, partial response, stable disease, progressive disease or not evaluable) since the start of treatment.
Time Frame: Tumor assessment was performed at screening and every 2nd course until earliest time of progression, death or end of treatment.
Population: Treated Set.
Measure: Number; unit: participants
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib | 400 mg Volasertib + 200 mg Nintedanib
Number analyzed (Participants) | 3 | 4 | 13 | 8 | 2
participants
  Complete Response | 0 | 0 | 1 | 0 | 0
  Partial Response | 0 | 0 | 1 | 0 | 0
  Stable Disease | 2 | 2 | 7 | 4 | 1
  Progressive Disease | 1 | 2 | 3 | 3 | 0
  Not Evaluable | 0 | 0 | 0 | 0 | 0
  Missing | 0 | 0 | 1 | 1 | 1

11. Secondary Outcome: Number of Patients With Objective Response (OR)
Description: Objective tumor response based on response evaluation criteria in solid tumors (RECIST) version 1.1. OR is defined as complete response (CR) or partial response (PR) as best response throughout the study.
Time Frame: as for outcome 10
Population: Treated Set.
Measure: Number; unit: participants
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib | 400 mg Volasertib + 200 mg Nintedanib
Number analyzed (Participants) | 3 | 4 | 13 | 8 | 2
participants
  Objective Response (OR) | 0 | 0 | 2 | 0 | 0
  Missing | 0 | 0 | 1 | 1 | 1

12. Primary Outcome: Maximum Tolerated Dose (MTD) of Volasertib in Combination With Nintedanib
Description: The MTD was determined using a 3+3 design with de-escalation. The MTD was defined as the highest dose level at which maximal 1 out of 6 patients experienced DLT in the first course of the escalation nd de-escalation phase. However, all DLT's occurring in the trial were considered for selection of the recommended dose for further development.
Time Frame: 28 days
Population: Treated Set. All patients who received >= 1 dose of study medication.
Measure: Number; unit: mg
Groups:
- Volasertib in Combination With Nintedanib: All patients received both Volasertib and Nintedanib. Starting dose of Volasertib was 100 mg, the next dose levels were 200 mg, 300 mg, 350 mg and 400 mg, which was to be infused on Day 8 in Course 1 and on Day 1 of subsequent courses. 200 mg Nintedanib was continuously administered twice daily except for the day of Volasertib administration.
Arm/Group | Volasertib in Combination With Nintedanib
Number analyzed (Participants) | 30
mg | 300

13. Secondary Outcome: Number of Patients With Disease Control
Description: Disease control based on response evaluation criteria in solid tumors (RECIST) version 1.1. Disease control is defined as complete response (CR), partial response (PR) or stable disease (SD) as best response throughout the study.
Time Frame: as for outcome 10
Population: Treated Set.
Measure: Number; unit: participants
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib | 400 mg Volasertib + 200 mg Nintedanib
Number analyzed (Participants) | 3 | 4 | 13 | 8 | 2
participants | 2 | 2 | 9 | 4 | 1

14. Secondary Outcome: Duration of Disease Control
Description: Disease control based on response evaluation criteria in solid tumors (RECIST) version 1.1. Patients who had a best overall tumour response of complete response (CR), partial response (PR) or stable disease (SD) were assessed to show disease control.
Time Frame: as for outcome 10
Population: All patients of the treated set that were assessed to show disease control.
Measure: Median (Full Range); unit: days
Groups:
- Total Patients: All patients received both Volasertib and Nintedanib. Volasertib was to be infused on Day 8 in Course 1 and on Day 1 of subsequent courses, dose level varied between 100mg and 400mg. 200 mg Nintedanib was continuously administered twice daily except for the day of Volasertib administration.
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib | 400 mg Volasertib + 200 mg Nintedanib | Total Patients
Number analyzed (Participants) | 2 | 2 | 9 | 4 | 1 | 18
days | 163.0 [114.0 to 212.0] | 348.0 [184.0 to 512.0] | 141.0 [74.0 to 447.0] | 215.0 [94.0 to 394.0] | 56.0 [56.0 to 56.0] | 161.5 [56.0 to 512.0]

15. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from start of treatment with study medication to tumour progression or death whichever occurs first. Tumour response was to be documented using appropriate techniques such as magnetic resonance imaging (MRI) or computer tomography (CT).
Time Frame: as for outcome 10
Population: Treated Set.
Measure: Median (Full Range); unit: days
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib | 400 mg Volasertib + 200 mg Nintedanib | Total Patients
Number analyzed (Participants) | 3 | 4 | 13 | 8 | 2 | 30
days | 114.0 [45.0 to 212.0] | 116.0 [35.0 to 512.0] | 99.0 [30.0 to 447.0] | 72.5 [8.0 to 394.0] | 83.0 [56.0 to 110.0] | 96.5 [8.0 to 512.0]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) that occurred during therapy with the study medication, or within 28 days after the last administration of any study medication, up to 485 days
Description: Patients were asked for spontaneous reports about AEs; detailed information was collected by specific questions.
Arm/Group | 100 mg Volasertib + 200 mg Nintedanib | 200 mg Volasertib + 200 mg Nintedanib | 300 mg Volasertib + 200 mg Nintedanib | 350 mg Volasertib + 200 mg Nintedanib | 400 mg Volasertib + 200 mg Nintedanib
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 5/13 | 2/8 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 13/13 | 8/8 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg Volasertib + 200 mg Nintedanib (N=3) | 200 mg Volasertib + 200 mg Nintedanib (N=4) | 300 mg Volasertib + 200 mg Nintedanib (N=13) | 350 mg Volasertib + 200 mg Nintedanib (N=8) | 400 mg Volasertib + 200 mg Nintedanib (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg Volasertib + 200 mg Nintedanib (N=3) | 200 mg Volasertib + 200 mg Nintedanib (N=4) | 300 mg Volasertib + 200 mg Nintedanib (N=13) | 350 mg Volasertib + 200 mg Nintedanib (N=8) | 400 mg Volasertib + 200 mg Nintedanib (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 9 | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 8 | 5 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0
Thyroid disorder (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3 | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 2 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 8 | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 2 | 4 | 6 | 1
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 6 | 3 | 2
Asthenia (General disorders) | 2 | 2 | 8 | 5 | 2
Chest pain (General disorders) | 3 | 1 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 2 | 2 | 0
Pyrexia (General disorders) | 0 | 1 | 5 | 4 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Viral uveitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 7 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 7 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 2 | 2 | 1
Glomerular filtration rate increased (Investigations) | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 2 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 3 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 2 | 2 | 1
Hypotension (Vascular disorders) | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.